CLINICAL TRIAL: NCT01351051
Title: A Multi-centre, Multinational, Cross-sectional, Incident Case-control Study on Factors Associated With the Development of Endometrioma and Deep Infiltrating Endometriosis
Brief Title: A Study of the Potential Risk Factors Linked to the Development of Severe Forms of Endometriosis
Acronym: FEELING
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-38-52014-185
Record Dates: First submitted 2011-04-08; First posted 2011-05-10 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- No endometriosis
- Superficial endometriosis
- Endometrioma
- Deep infiltrating endometriosis

SUMMARY:
This study will aim to identify genetic, medical, dietary and environmental factors associated with the development of endometrioma and/or deep infiltrating endometriosis in order to move towards early diagnosis and implementation of potential preventative measures.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a female aged between 18 and 41 years
* The subject has undergone a laparoscopy or laparotomy for a benign gynecological indication excluding pregnancy, in the last 3 months
* The subject's surgery showed either no visible endometriosis lesions or histologically confirmed endometriosis lesions: superficial endometriosis, endometrioma or deep infiltrating endometriosis
* The subject has given a written informed consent prior to any study-related procedures

Exclusion Criteria:

* The subject is pregnant
* The subject's surgery results showed evidence of malignancy
* The subject has a mental condition rendering her unable to understand the nature, scope and possible consequences of the study, and/or with evidence of an uncooperative attitude

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who have undergone a laparoscopy/laparatomy for a benign gynaecological indication excluding pregnancy in the last 3 months.
Sampling Method: Probability Sample
Enrollment: 1008 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Factors associated with endometrioma and/or deep infiltrating endometriosis using retrospective data collection and patient questionnaire. | Enrolment visit

SECONDARY OUTCOMES:
Factors associated with superficial endometriosis using retrospective data collection and patient questionnaire. | Enrolment visit
Factors associated with endometrioma and/or deep infiltrating endometriosis according to subject ethnicity using retrospective data collection and patient questionnaire. | Enrolment visit
Subject's characteristics by endometriosis status using retrospective data collection and patient questionnaire. | Enrolment visit

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (7):
- China (4):
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - The Third Xiangya Hospital of Central South University, Changsha
  - Women's Hospital School of Medicine, Zhejiang University, Zhejiang
- Hôpital St Vincent de Paul, Paris, France
- Russia (2):
  - Research Institute of Maternity and Childhood named after V.N. Gorodkov, Ivanovo
  - Moscow Regional Scientific Research Institute of Obstetrics and Gynaecology, Moscow

REFERENCES:
- [Derived] Dai Y, Zhou Y, Zhang X, Xue M, Sun P, Leng J, Chapron C. Factors associated with deep infiltrating endometriosis versus ovarian endometrioma in China: a subgroup analysis from the FEELING study. BMC Womens Health. 2018 Dec 22;18(1):205. doi: 10.1186/s12905-018-0697-7. PMID 30577792
- [Derived] Chapron C, Lang JH, Leng JH, Zhou Y, Zhang X, Xue M, Popov A, Romanov V, Maisonobe P, Cabri P. Factors and Regional Differences Associated with Endometriosis: A Multi-Country, Case-Control Study. Adv Ther. 2016 Aug;33(8):1385-407. doi: 10.1007/s12325-016-0366-x. Epub 2016 Jun 24. PMID 27342743